CLINICAL TRIAL: NCT02933398
Title: A Prospective Randomized Controlled Trial Comparing Two Minimally Invasive Surgical Modalities - Robotic Assisted Vs. Pure Laparoscopic Partial Nephrectomy For Small Renal Masses.
Brief Title: A Trial Comparing - Robotic Assisted Versus Laparoscopic Partial Nephrectomy For Small Renal Masses
Acronym: RALPLPNNX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RALPLPNNX
Record Dates: First submitted 2014-10-10; First posted 2016-10-14 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Small Renal Masses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Assisted Partial Nephrectomy (Active Comparator): Current standard for partial nephrectomies.
  Interventions: Procedure: Robotic Assisted Nephrectomy
- Robotic Assisted Partial Nephrectomy (Active Comparator): Possible new standard for partial nephrectomies.
  Interventions: Procedure: Laparoscopic Assisted Nephrectomy

INTERVENTIONS:
Procedure: Robotic Assisted Nephrectomy — Robotic (Davinci)
  Arms: Laparoscopic Assisted Partial Nephrectomy
Procedure: Laparoscopic Assisted Nephrectomy — Regular Laparoscopic Technique.
  Arms: Robotic Assisted Partial Nephrectomy

SUMMARY:
A prospective, randomized, controlled trial including patients who are diagnosed with a small renal mass (<4 cm) amenable to resection using either RALPN or LPN.

DETAILED DESCRIPTION:
Small renal masses (SRM) <4cm are increasingly being discovered incidentally on imaging. The standard of care for management of SRMs is partial nephrectomy whenever feasible. In the last 10 years, a minimally invasive laproscopic approach has largely supplanted open surgery for the treatment of SRMs. Robot-assisted laparoscopic partial nephrectomy (RALPN) has emerged as an alternative to laparoscopic partial nephrectomy (LPN) and has been able to bridge the technical difficulties of LPN. The big question about the role and cost of RALPN in comparison to LPN especially in Canadian healthcare for SRMs still remains unanswered.

The objective of this proposed study is to conduct a randomized controlled trial to determine whether RALPN is better than LPN for the management of patients with SRMs. The primary outcomes will be warm ischemia time and secondary outcomes will be estimated glomerular filtration rate (eGFR), estimated blood loss, complication rate, length of hospital stay, positive surgical margin rate and cost comparison of these two techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years of age and capable of giving informed consent
2. Patients scheduled for treatment of a renal tumor suitable to undergo LPN /RALPN
3. Patients with SRMs (tumor(s) ≤ 4 cm)

Exclusion Criteria:

1. Large tumors > 4.0cm
2. Unable to have a general anesthetic
3. Unable to comply with post-operative follow-up protocol
4. Uncorrectable bleeding diathesis
5. Tumors unsuitable for LPN/RALPN technique
6. Evidence of metastatic disease
7. Prior surgery on the affected kidney
8. Ectopic or malrotated kidney
9. Mental health condition that precludes informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Warm ischemia time | Duration of the Surgical Procedure (Nephrectomy)
  It will be measured intraoperatively from the time of application of Satinsky clamp on the renal hilum to the release of clamp (in minutes).

SECONDARY OUTCOMES:
eGFR | Up to 24 months post operatively.
  It will be measured preoperatively, postoperatively and at each of the follow-up visit.
Estimated blood loss | Duration of the Surgical Procedure (Nephrectomy)
  Will be measured intraoperatively from the amount of blood (ml) in the suction container.
Complication rates as per Clavien-Dindo classification | Up to 24 months post-operatively.
  It will be recorded for the intra-operative, post-operative and follow-up period.
Conversion rate to radical nephrectomy or OPN due to technical difficulty. | Duration of the Surgical Procedure
  From the start of the partial nephrectomy in minutes to the time it was decided to convert to a radical nephrectomy.
Postoperative pain | Minutes to hours after nephrectomy up to 3 months post-operatively.
Length of hospital stay | 3-7 Days
  Calculated from day of admission to day of discharge from hospital.
Positive surgical margin rate | 14 days
  Will be based on the final pathology results which are usually ready in 1-2 weeks post surgery. Distance to surgical margin will be looked at (mm to cm).
Costs of treatment | Up to 1 year
  Clinical data and resource use for both treatments will be collected and unit cost estimates will be based on the St. Joseph Healthcare case-costing system. The cost will be conducted from the perspective of Ontario Ministry of Health and Long-term Care. The cost of hospital stay will be calculated along with any hospital stay/procedure associated with a post-op complication.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton - McMaster Institute of Urology, Hamilton, Ontario, Canada